CLINICAL TRIAL: NCT06525389
Title: Liposomal Amphotericin B and Flucytosine Antifungal Strategy for Talaromycosis (LAmB-FAST)
Acronym: LAmB-FAST
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Pham Ngoc Thach University of Medicine (Other); Hospital for Tropical Diseases, Ho Chi Minh City, Vietnam (Other); National Hospital for Tropical Diseases, Hanoi, Vietnam (Other Government); Bach Mai Hospital (Other); Gilead Sciences (Industry); Viatris Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00113856
Record Dates: First submitted 2024-07-24; First posted 2024-07-29 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-04

CONDITIONS: Talaromycosis
Keywords: Penicilliosis; Talaromyces marneffei infection; Penicillium marneffei infection
MeSH Terms: conditions — talaromycosis | interventions — liposomal amphotericin B; Flucytosine; amphotericin B, deoxycholate drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Liposomal amphotericin B vs deoxycholate amphotericin B arm is an open label comparison
  Flucytosine vs no flucytosine is a placebo controlled comparison
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Deoxycholate Amphotericin B (DAmB) plus Flucytosine (5FC) placebo (Active Comparator): DAmB (0.7mg/kg/d IV x 14 days) + 5FC placebo (25 mg/kg oral 3x daily x 14 days)
  Interventions: Drug: Flucytosine (5FC) placebo pill; Drug: Deoxycholate Amphotericin B (DAmB)
- Deoxycholate Amphotericin B (DAmB) plus Flucytosine (5FC) (Experimental): DAmB (0.7 mg/kg/d IV x 14 days) + 5FC (25 mg/kg oral 3x daily x 14 days)
  Interventions: Drug: Flucytosine (5FC); Drug: Deoxycholate Amphotericin B (DAmB)
- Liposomal Amphotericin B (LAmB) plus Flucytosine (5FC) placebo (Experimental): LAmB (10 mg/kg IV x 1 dose) + 5FC placebo (25 mg/kg oral 3x daily x 14 days)
  Interventions: Drug: Liposomal Amphotericin B (LAmB); Drug: Flucytosine (5FC) placebo pill
- Liposomal Amphotericin B (LAmB) plus Flucytosine (5FC) (Experimental): LAmB (10 mg/kg IV x 1 dose) + 5FC (25 mg/kg oral 3x daily x 14 days)
  Interventions: Drug: Liposomal Amphotericin B (LAmB); Drug: Flucytosine (5FC)

INTERVENTIONS:
Drug: Liposomal Amphotericin B (LAmB) — Antifungal dosed at 10 mg/kg/day IV x one single dose.
  Arms: Liposomal Amphotericin B (LAmB) plus Flucytosine (5FC); Liposomal Amphotericin B (LAmB) plus Flucytosine (5FC) placebo
Drug: Flucytosine (5FC) — Antifungal dosed at 25mg/kg oral 3x daily.
  Arms: Deoxycholate Amphotericin B (DAmB) plus Flucytosine (5FC); Liposomal Amphotericin B (LAmB) plus Flucytosine (5FC)
Drug: Flucytosine (5FC) placebo pill — Similar in appearance to flucytosine. Also dosed at 25mg/kg oral 3x daily.
  Arms: Deoxycholate Amphotericin B (DAmB) plus Flucytosine (5FC) placebo; Liposomal Amphotericin B (LAmB) plus Flucytosine (5FC) placebo
Drug: Deoxycholate Amphotericin B (DAmB) — Antifungal dosed at 0.7 mg/kg/day IV x 2 weeks.
  Arms: Deoxycholate Amphotericin B (DAmB) plus Flucytosine (5FC); Deoxycholate Amphotericin B (DAmB) plus Flucytosine (5FC) placebo

SUMMARY:
LAmB-FAST is a factorial randomized controlled trial simultaneously testing two interventions in one trial. LAmB-FAST seeks to inform treatment guidelines on the induction and maintenance therapy of HIV-associated talaromycosis (formerly called penicilliosis) and will answer the following three questions:

1. Is induction therapy using a single 10 mg\/kg dose of liposomal amphotericin B (LAmB) is more effective than 14 days of the conventional deoxycholate amphotericin B (DAmB)?
2. Is adding flucytosine (5FC) to amphotericin B more effective than amphotericin B alone?
3. Is HIV viral load guided stopping of itraconazole maintenance therapy as effective as the current CD4 guided strategy in the prevention of talaromycosis relapse?

DETAILED DESCRIPTION:
Talaromycosis (formerly known as penicilliosis) is caused by the dimorphic fungus Talaromyces marneffei (Tm) endemic in Southeast Asia where it is a leading the cause of death among people with advanced HIV disease (AHD, CD4 count <200 cells/mm3 and/or WHO disease stage III or IV). Despite the mortality on treatment as high as 30%, current treatment options are limited to just two drugs: amphotericin B deoxycholate (DAmB) - which has substantial toxicity, and itraconazole - which has poor bioavailability.

As a roadmap to identify safer and more effective antifungal strategies, LAmB-FAST applies major advances made in HIV-associated mycoses to accelerate treatment for HIV-associated talaromycosis. First, clinical trials in cryptococcosis showed that shorter courses (5 to 7 days) of DAmB was as effective and less toxic than the standard 14-day course of DAmB. The recent AMBITION cryptococcal meningitis showed that a single 10 mg/kg dose of liposomal amphotericin B (LAmB) was as effective as 7 to 14 days of DAmB but had 30% less toxicity, leading to rapid endorsement by the WHO as the first-line therapy for cryptococcal meningitis in 2022. A single LAmB induction therapy strategy has also been demonstrated in a phase II HIV-associated histoplasmosis trial which showed that a single 10 mg/kg dose of LAmB had similar mortality compared to 2 doses or 14 daily doses of LAmB. Second, the addition of flucytosine (5FC) to DAmB has been shown to improves fungal clearance in the cerebrospinnal fluid and survival of patients with cryptococcal meningitis. These advances in other HIV-associated mycoses lead us to hypothesize that 1) a single 10mg/kg dose of LAmB will be superior to 14 days of DAmB and 2) the addition of 5FC will be superior to DAmB or LAmB alone in the induction therapy of talaromyosis.

LAmB-FAST will test three related but independent specific aims: AIM 1: To determine if a single 10mg/kg dose of LAmB is superior to 14 days of DAmB in Tm complication-free survival. AIM 2:

To determine if combination therapy with 5FC is superior to DAmB or LAmB alone in Tm complication-free survival.

The primary outcome (for both AIM 1 and AIM 2) is hazard of a composite of death, Tm complications, and adverse events (AEs) grade 3 or higher.

The secondary outcomes include:

1. All-cause mortality;
2. Fungal clearance rate over first 14 days;
3. A novel 4-scale hierarchical outcome of i. Mortality, ii. Tm complications, iii. AEs grade 3, iv. Quality of life scores;
4. Rates of Tm DNA and Tm antigen decline over first 12 weeks.

AIM 3 will leverage access to a well-characterized and treated talaromycosis cohort in AIM 1 and AIM 2 to conduct a follow-on nested randomized controlled sub-study testing whether a HIV viral load guided strategy of stopping itraconazole chemoprophylaxis (STOP SHORT) is non-inferior to the current CD4 guided strategy in the prevention of talaromycosis relapse and death.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected adults (age greater or equal to 18), on ART or no ART
* Definitive talaromycosis confirmed by microscopy, histology, or culture

Exclusion Criteria:

* Known severe allergy to AmB or 5FC
* Absolute neutrophil count <500 cells
* Concurrent cryptococcal or TB meningitis
* Received > 2 doses of DAmB
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 428 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2030-11-01 (Estimated); Study Completion 2031-11-01 (Estimated)

PRIMARY OUTCOMES:
Time from enrollment to a composite of poor outcomes | up to 24 weeks
  Poor outcomes are defined as of death, talaromycosis complications (defined as relapse, immune inflammatory reconstitution inflammatory syndrome [IRIS], wasting syndrome [>10% weight loss from enrollment], re-hospitalization, and grade 3 or higher adverse events

SECONDARY OUTCOMES:
All cause mortality | up to 24 weeks
Fungal clearance rate as measured by early fungicidal activity (EFA) in log10 CFUs/mL/day | 14 days
Composite ordinal desirability of outcome ranking (DOOR) scale | over 24 weeks
  All-cause mortality, Talaromycosis complications and adverse events grade 4, Adverse events grade 3, and Quality of Life (QOL) utility scores by EQ5D scale.
Change in Talaromyces marneffei DNA in copies/mL/week | baseline to 24 weeks
Change in Talaromyces marneffei antigen in µg/mL/week | baseline to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Thuy Le, MD, PhD, Principal Investigator — Duke University
Locations (5):
- Duke University Medical Center, Durham, North Carolina, United States
- Vietnam (4):
  - Bach Mai Hospital, Hanoi
  - National Hospital for Tropical Diseases, Hanoi
  - Hospital for Tropical Diseases, Ho Chi Minh City
  - Pham Ngoc Thach University of Medicine, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Data sharing with the scientific community will be carried out according to the FAIR Guiding Principles and spirit of open-access. Previously published data sets will be made available to the scientific community upon request after agreement by the Trial Steering Commitee. The Duke Data Manager will deposit the de-identified master data file into the Duke Research Data Repository (RDR), an openly accessible preservation archive maintained by the Duke University Libraries.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will become available when all primary and secondary analyses are completed and published and will be available in the Duke Research Data Repository (RDR) indefinitely
Access Criteria: Contact PI